CLINICAL TRIAL: NCT01281306
Title: A Multi-center, Randomized, Double-blind, Placebo and Active Controlled, Parallel Group Study to Evaluate the Dose Response of AHU377 in Combination With Valsartan 320 mg After 8 Week Treatment in Patients With Mild-to-moderate Systolic Hypertension
Brief Title: An 8-week Study to Evaluate the Dose Response of AHU377 in Combination With Valsartan 320 mg in Patients With Mild-to-moderate Systolic Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLCZ696A2223; 2010-022326-32
Record Dates: First submitted 2011-01-20; First posted 2011-01-21 (Estimated); Results first posted 2015-08-18 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2015-12

CONDITIONS: Systolic Hypertension
Keywords: hypertension; blood pressure; LCZ696; dual-acting; neprilysin; nep inhibitor; vasopeptidase; angiotensin receptor; angiotensin receptor neprilysin inhibitor (ARNi)
MeSH Terms: conditions — Isolated Systolic Hypertension; Hypertension | interventions — sacubitril and valsartan sodium hydrate drug combination; Valsartan; sacubitril

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (7):
- VAL + AHU 400 mg (Experimental): Participants were started with AHU377 100 mg + valsartan 160 mg every day (qd) for 1 week, then were uptitrated to AHU377 200 mg + valsartan 320 mg qd for another week, and then were uptitrated to AHU377 400 mg + valsartan 320 mg for the remaining 6 weeks.
  Interventions: Drug: Valsartan; Drug: AHU377
- VAL + AHU 200 mg (Experimental): Participants were started with AHU377 100 mg + valsartan 160 mg qd for 1 week and then were uptitrated to AHU377 200 mg + valsartan 320 mg qd for the remaining 7 weeks.
  Interventions: Drug: Valsartan; Drug: AHU377
- VAL + AHU 100 mg (Experimental): Participants were started with AHU377 50 mg + valsartan 160 mg qd for 1 week and then were uptitrated to AHU377 100 mg + valsartan 320 mg for the remaining 7 weeks.
  Interventions: Drug: Valsartan; Drug: AHU377
- VAL + AHU 50 mg (Experimental): Participants were started with AHU377 50 mg + valsartan 160 mg qd for 1 week and then were uptitrated to AHU377 50 mg + valartan 320 mg qd for the remaining 7 weeks.
  Interventions: Drug: Valsartan; Drug: AHU377
- VAL 320 mg (Experimental): Participants were started with valsartan 160 mg qd for 1 week and then were uptitrated to valsartan 320 mg qd for the remaining 7 weeks.
  Interventions: Drug: Valsartan
- LCZ 400 mg (Experimental): Participants were started with LCZ696 200 mg qd for 1 week and then were uptitrated to LCZ696 400 mg qd for the remaining 7 weeks.
  Interventions: Drug: LCZ696
- Placebo (Experimental): Participants received matching placebo to LCZ696, AHU377 and valsartan for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LCZ696 — LCZ696 was supplied as tablets in blister cards in 100 mg strengths.
  Arms: LCZ 400 mg
Drug: Valsartan — Valsartan was supplied as tablets in blister cards in 160 mg and 320 mg strengths.
  Arms: VAL + AHU 100 mg; VAL + AHU 200 mg; VAL + AHU 400 mg; VAL + AHU 50 mg; VAL 320 mg
Drug: AHU377 — AHU377 was supplied in tablets in blister cards in 50 mg and 100 mg strengths.
  Arms: VAL + AHU 100 mg; VAL + AHU 200 mg; VAL + AHU 400 mg; VAL + AHU 50 mg
Drug: Placebo — Placebo was supplied as tablets in blister cards.
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate dose response of blood pressure lowering for 4 doses of AHU377, given once daily (50 mg, 100 mg, 200 mg and 400 mg) in combination with a fixed dose of valsartan (320 mg).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed. Patients with mild-to-moderate systolic hypertension, untreated or currently taking antihypertensive therapy.
* Ability to communicate and comply with all study requirements and demonstrate good medication compliance (≥ 80% compliance rate) during the run-in period.

Exclusion Criteria:

* Severe hypertension
* History of angioedema, drug-related or otherwise, as reported by the patient.
* Pregnant or nursing (lactating) women.
* Women of child-bearing potential (WOCBP), UNLESS they are using adequate birth control methods.
* History or evidence of a secondary form of hypertension.
* Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 910 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (74):
- United States (15):
  - Novartis Investigative Site, Clearwater, Florida
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Metairie, Louisiana
  - Novartis Investigative Site, Belzoni, Mississippi
  - Novartis Investigative Site, Jackson, Mississippi
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Henderson, Nevada
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Buffalo, New York
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Greensboro, North Carolina
  - Novartis Investigative Site, Shelby, North Carolina
  - Novartis Investigative Site, Erie, Pennsylvania
  - Novartis Investigative Site, Bryan, Texas
  - Novartis Investigative Site, Houston, Texas
- Argentina (8):
  - Novartis Investigative Site, Buenos Aires, Buenos Aires
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, Lanús, Buenos Aires
  - Novartis Investigative Site, Caba, Buenos Aires F.D.
  - Novartis Investigative Site, Corrientes, Corrientes Province
  - Novartis Investigative Site, Córdoba, Córdoba Province
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
- Canada (3):
  - Novartis Investigative Site, Mount Pearl, Newfoundland and Labrador
  - Novartis Investigative Site, Mirabel, Quebec
  - Novartis Investigative Site, Ste-Foy, Quebec
- Hungary (7):
  - Novartis Investigative Site, Csongrád, Hungary
  - Novartis Investigative Site, Érd, Hungary
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Miskolc
  - Novartis Investigative Site, Nyiregyháza
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Törökbálint
- India (7):
  - Novartis Investigative Site, Visakhapatnam, Andhra Pradesh
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Nashik, Maharashtra
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, Ludhiana, Punjab
  - Novartis Investigative Site, Jaipur, Rajasthan
  - Novartis Investigative Site, Lucknow, Uttar Pradesh
- Romania (5):
  - Novartis Investigative Site, Bucharest, District 1
  - Novartis Investigative Site, Bucharest, District 2
  - Novartis Investigative Site, Oradea, Jud. Bihor
  - Novartis Investigative Site, Craiova, Jud. Dolj
  - Novartis Investigative Site, Bucharest
- Slovakia (12):
  - Novartis Investigative Site, Nitra, Slovak Republic
  - Novartis Investigative Site, Prešov, Slovak Republic
  - Novartis Investigative Site, Bratislava, Slovakia
  - Novartis Investigative Site, Liptovský Mikuláš, Slovakia
  - Novartis Investigative Site, Nitra, Slovakia
  - Novartis Investigative Site, Nové Zámky, Slovakia
  - Novartis Investigative Site, Partizánske, Slovakia
  - Novartis Investigative Site, Prešov, Slovakia
  - Novartis Investigative Site, Ružomberok, Slovakia
  - Novartis Investigative Site, Sereď, Slovakia
  - Novartis Investigative Site, Šaľa, Slovakia
  - Novartis Investigative Site, Zvolen, Slovakia
- South Korea (7):
  - Novartis Investigative Site, Bucheon-si, Gyeonggi-do
  - Novartis Investigative Site, Goyang-si, Gyeonggi-do
  - Novartis Investigative Site, Uijeongbu-si, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Koyang, Kyunggi
  - Novartis Investigative Site, Seoul, Seoul
  - Novartis Investigative Site, Seoul
- Spain (10):
  - Novartis Investigative Site, Granada, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Centelles, Catalonia
  - Novartis Investigative Site, Tarragona, Catalonia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Alzira, Valencia
  - Novartis Investigative Site, Barcelona

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study consisted of a single-blind run-in period and a double-blind (DB) period. During the 3 to 4 week run-in, participants were assessed for randomization eligibility into the DB period. 910 participants randomized. 3 participants were mis-randomized and did not receive study treatment. Therefore, the participant flow shows 907 participants.
Pre-assignment Details: In the double blind period, participants were randomized in a 2:2:2:2:2:2:1 ratio to AHU377 400 mg + valsartan 320 mg, AHU377 200 mg + valsartan 320 mg, AHU377 100 mg + valsartan 320 mg, AHU377 50 mg + valsartan 320 mg,valsartan 320 mg, LCZ696 400 mg and placebo, respectively.
Period: Overall Study
Arm/Group | VAL + AHU 400 mg | VAL + AHU 200 mg | VAL + AHU 100 mg | VAL + AHU 50 mg | VAL 320 mg | LCZ 400 mg | Placebo
Started | 144 | 145 | 141 | 134 | 143 | 142 | 58
Full Analysis Set | 143 | 145 | 141 | 133 | 143 | 142 | 58
Safety Set | 143 | 145 | 141 | 133 | 143 | 142 | 58
Ambulatory Blood Pressure Monitoring Set | 95 | 99 | 92 | 95 | 93 | 91 | 35
Completed | 136 | 141 | 133 | 123 | 134 | 135 | 51
Not Completed | 8 | 4 | 8 | 11 | 9 | 7 | 7
Not completed — Lack of Efficacy | 0 | 1 | 3 | 0 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 2 | 4 | 1 | 3 | 1
Not completed — Protocol deviation | 0 | 1 | 1 | 1 | 1 | 0 | 0
Not completed — Condition no longer requires study drug | 1 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 2 | 0 | 0 | 1
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 2 | 2 | 3 | 5 | 3 | 3
Not completed — Randomized in error | 1 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VAL + AHU 400 mg | VAL + AHU 200 mg | VAL + AHU 100 mg | VAL + AHU 50 mg | VAL 320 mg | LCZ 400 mg | Placebo | Total
Number analyzed (Participants) | 144 | 145 | 141 | 134 | 143 | 142 | 58 | 907
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.7 (11.36) | 61.7 (11.44) | 61.0 (11.03) | 62.0 (10.73) | 62.0 (11.45) | 61.2 (10.60) | 60.8 (11.81) | 61.5 (11.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 60 | 53 | 61 | 60 | 71 | 29 | 412
  Male | 66 | 85 | 88 | 73 | 83 | 71 | 29 | 495

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure (msSBP)
Description: Sitting BP measurements were performed at trough (23-26 hours post-morning dose). A negative change from baseline indicates improvement.
Time Frame: Baseline, 8 weeks
Population: Only participants of the full analysuis set (FAS), who had measurements at both baseline and week 8, were included in the analysis. The FAS included all randomized participants who received at least one dose of double-blind study medication.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | VAL + AHU 400 mg | VAL + AHU 200 mg | VAL + AHU 100 mg | VAL + AHU 50 mg | VAL 320 mg | LCZ 400 mg | Placebo
Number analyzed (Participants) | 143 | 144 | 141 | 132 | 143 | 142 | 57
mmHg | -20.89 (1.22) | -23.55 (1.21) | -21.26 (1.23) | -19.31 (1.27) | -16.13 (1.22) | -21.78 (1.22) | -6.99 (1.92)

2. Secondary Outcome: Change From Baseline in Mean Diastolic Blood Pressure (msDBP)
Description: as for outcome 1
Time Frame: Baseline, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | VAL + AHU 400 mg | VAL + AHU 200 mg | VAL + AHU 100 mg | VAL + AHU 50 mg | VAL 320 mg | LCZ 400 mg | Placebo
Number analyzed (Participants) | 143 | 144 | 141 | 132 | 143 | 142 | 57
mmHg | -8.47 (0.76) | -9.76 (0.75) | -8.04 (0.76) | -7.15 (0.79) | -7.28 (0.76) | -9.61 (0.75) | -3.38 (1.19)

3. Secondary Outcome: Change From Baseline in Mean 24 Hour Ambulatory SBP (maSBP) and Mean 24 Hour Ambulatory DBP (maDBP)
Description: Twenty four hour ABPM was performed twice duirng the study at baseline and week 8. The second ABPM assessment was performed only in participants who had successfully completed the ABPM assessment at baseline. A negative change from baseline indicates improvement.
Time Frame: Baseline, 8 weeks
Population: A subset of randomized participants, who had ABPM measurements at both baseline and week 8, were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | VAL + AHU 400 mg | VAL + AHU 200 mg | VAL + AHU 100 mg | VAL + AHU 50 mg | VAL 320 mg | LCZ 400 mg | Placebo
Number analyzed (Participants) | 94 | 98 | 92 | 95 | 93 | 90 | 35
mmHg
  maSBP | -12.14 (0.71) | -15.66 (0.69) | -14.33 (0.72) | -11.36 (0.70) | -9.59 (0.71) | -12.98 (0.71) | -2.12 (1.15)
  maDBP | -5.81 (0.44) | -7.03 (0.42) | -6.46 (0.44) | -5.36 (0.43) | -5.23 (0.44) | -6.20 (0.44) | -0.79 (0.71)

4. Secondary Outcome: Change From Baseline in Daytime maSBP and maDBP
Description: Twenty four hour ABPM was performed twice during the study at baseline and week 8. The second ABPM assessment was performed only in participants who had successfully completed the ABPM assessment at baseline. A negative change from baseline indicates improvement.
Time Frame: Baseline, 8 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | VAL + AHU 400 mg | VAL + AHU 200 mg | VAL + AHU 100 mg | VAL + AHU 50 mg | VAL 320 mg | LCZ 400 mg | Placebo
Number analyzed (Participants) | 94 | 98 | 92 | 95 | 93 | 90 | 35
mmHg
  maSBP | -12.62 (1.21) | -15.85 (1.19) | -14.43 (1.23) | -11.50 (1.21) | -9.60 (1.22) | -13.32 (1.23) | -2.39 (1.98)
  maDBP | -5.93 (0.77) | -7.13 (0.75) | -6.57 (0.78) | -5.39 (0.77) | -5.40 (0.77) | -6.16 (0.78) | -0.98 (1.26)

5. Secondary Outcome: Change From Baseline in Nighttime maSBP and maDBP
Description: as for outcome 3
Time Frame: Baseline and 8 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | VAL + AHU 400 mg | VAL + AHU 200 mg | VAL + AHU 100 mg | VAL + AHU 50 mg | VAL 320 mg | LCZ 400 mg | Placebo
Number analyzed (Participants) | 91 | 98 | 90 | 95 | 92 | 90 | 35
mmHg
  maSBP | -11.57 (1.23) | -15.27 (1.19) | -14.74 (1.23) | -10.80 (1.21) | -8.88 (1.22) | -12.34 (1.23) | -1.36 (1.98)
  maDBP | -5.27 (0.78) | -6.79 (0.75) | -6.45 (0.78) | -5.27 (0.77) | -4.49 (0.77) | -6.36 (0.78) | -0.22 (1.26)

6. Secondary Outcome: Change From Baseline in Mean Sitting Pulse Pressure
Description: Pulse rate measurements were performed. A negative change from baseline indicates improvement.
Time Frame: Baseline, 8 weeks
Population: Only participants of the full analysis set (FAS), who had measurements at both baseline and week 8, were included in the analysis. The FAS included all randomized participants who received at least one dose of double-blind study medication.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | VAL + AHU 400 mg | VAL + AHU 200 mg | VAL + AHU 100 mg | VAL + AHU 50 mg | VAL 320 mg | LCZ 400 mg | Placebo
Number analyzed (Participants) | 143 | 144 | 141 | 132 | 143 | 142 | 57
mmHg | -12.39 (0.91) | -13.91 (0.90) | -13.18 (0.91) | -12.01 (0.95) | -8.80 (0.91) | -12.18 (0.91) | -3.74 (1.43)

7. Secondary Outcome: Change From Baseline in Mean Ambulatory Pulse Pressure
Description: Pulse rate measurements were performed. A negative change from baseline indicates improvement.
Time Frame: Baseline, 8 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | VAL + AHU 400 mg | VAL + AHU 200 mg | VAL + AHU 100 mg | VAL + AHU 50 mg | VAL 320 mg | LCZ 400 mg | Placebo
Number analyzed (Participants) | 94 | 98 | 92 | 95 | 93 | 90 | 35
mmHg | -6.23 (0.39) | -8.51 (0.38) | -7.71 (0.40) | -6.00 (0.39) | -4.40 (0.39) | -6.84 (0.39) | -1.09 (0.63)

8. Secondary Outcome: Change From Baseline in maSBP and maDBP in Dippers
Description: Twenty four hour ABPM was performed twice during the study at baseline and week 8. The second ABPM assessment was performed only in participants who had successfully completed the ABPM assessment at baseline. Dippers were defined as participants who showed a decrease of at least 10% in maSBP during the night (10pm-6am) compared with the daytime level. A negative change from baseline indicates improvement.
Time Frame: Baseline, 8 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | VAL + AHU 400 mg | VAL + AHU 200 mg | VAL + AHU 100 mg | VAL + AHU 50 mg | VAL 320 mg | LCZ 400 mg | Placebo
Number analyzed (Participants) | 32 | 42 | 38 | 42 | 38 | 37 | 19
mmHg
  maSBP | -11.43 (1.12) | -15.59 (1.00) | -12.04 (1.05) | 10.60 (1.01) | -9.85 (1.03) | -13.09 (1.05) | -2.39 (1.45)
  maDBP | -4.62 (0.70) | -7.33 (0.62) | -5.49 (0.65) | -5.07 (0.63) | -5.53 (0.64) | -6.03 (0.65) | -0.98 (0.90)

9. Secondary Outcome: Change From Baseline in maSBP and maDBP in Non-dippers
Description: Twenty four hour ABPM was performed twice duirng the study at baseline and week 8. The second ABPM assessment was performed only in participants who had successfully completed the ABPM assessment at baseline. Dippers were defined as participants who showed a decrease of at least 10% in maSBP during the night (10pm-6am) compared with the daytime level. A negative change from baseline indicates improvement.
Time Frame: Baseline, 8 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | VAL + AHU 400 mg | VAL + AHU 200 mg | VAL + AHU 100 mg | VAL + AHU 50 mg | VAL 320 mg | LCZ 400 mg | Placebo
Number analyzed (Participants) | 59 | 56 | 53 | 53 | 54 | 53 | 16
mmHg
  maSBP | -12.81 (0.91) | -16.08 (0.94) | -16.37 (0.97) | -12.17 (0.99) | -9.73 (0.96) | -13.12 (0.96) | -1.46 (1.75)
  maDBP | -6.65 (0.56) | -6.91 (0.58) | -7.31 (0.60) | -5.79 (0.61) | -5.10 (0.59) | -6.34 (0.59) | -0.49 (1.08)

10. Secondary Outcome: Change From Baseline in msSBP and msDBP in Participants < 65 Years of Age
Description: as for outcome 1
Time Frame: Baseline, 8 weeks
Population: Only participants of the full analysuis set (FAS), who were < 65 years of age and had measurements at both baseline and week 8, were included in the analysis. The FAS included all randomized participants who received at least one dose of double-blind study medication.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | VAL + AHU 400 mg | VAL + AHU 200 mg | VAL + AHU 100 mg | VAL + AHU 50 mg | VAL 320 mg | LCZ 400 mg | Placebo
Number analyzed (Participants) | 75 | 75 | 78 | 66 | 73 | 79 | 28
mmHg
  msSBP | -20.95 (1.68) | -24.45 (1.67) | -20.94 (1.63) | -18.09 (1.79) | -16.96 (1.71) | -21.06 (1.63) | -8.94 (2.73)
  msDBP | -8.97 (1.11) | -10.94 (1.11) | -8.83 (1.09) | -8.07 (1.19) | -6.93 (1.13) | -10.25 (1.08) | -5.19 (1.82)

11. Secondary Outcome: Change From Baseline in msSBP and msDBP in Participants >= 65 Years of Age
Description: as for outcome 1
Time Frame: Baseline, 8 weeks
Population: Only participants of the full analysuis set (FAS), who were >= 65 years of age and had measurements at both baseline and week 8, were included in the analysis. The FAS included all randomized participants who received at least one dose of double-blind study medication.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | VAL + AHU 400 mg | VAL + AHU 200 mg | VAL + AHU 100 mg | VAL + AHU 50 mg | VAL 320 mg | LCZ 400 mg | Placebo
Number analyzed (Participants) | 68 | 69 | 63 | 66 | 70 | 63 | 29
mmHg
  msSBP | -20.93 (1.79) | -22.66 (1.76) | -21.72 (1.85) | -20.64 (1.81) | -15.48 (1.75) | -22.83 (1.84) | -5.10 (2.71)
  msDBP | -7.89 (1.02) | -8.44 (1.00) | -7.06 (1.05) | -6.17 (1.03) | -7.62 (0.99) | -8.89 (1.04) | -1.46 (1.54)

12. Secondary Outcome: Change From Baseline in maSBP and maDBP in Participants < 65 Years of Age
Description: as for outcome 3
Time Frame: Baseline, 8 weeks
Population: A subset of randomized participants, who were leass than 65 years of age and had ABPM measurements at both baseline and week 8, were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | VAL + AHU 400 mg | VAL + AHU 200 mg | VAL + AHU 100 mg | VAL + AHU 50 mg | VAL 320 mg | LCZ 400 mg | Placebo
Number analyzed (Participants) | 44 | 50 | 46 | 47 | 44 | 48 | 15
mmHg
  maSBP | -12.16 (0.98) | -15.06 (0.91) | -14.42 (0.95) | -10.39 (0.95) | -9.55 (0.99) | -13.98 (0.93) | -2.24 (1.67)
  maDBP | -6.74 (0.67) | -7.81 (0.62) | -7.93 (0.65) | -5.69 (0.65) | -5.94 (0.67) | -7.32 (0.63) | -1.53 (1.14)

13. Secondary Outcome: Change From Baseline in maSBP and maDBP in Participants >= 65 Years of Age
Description: as for outcome 3
Time Frame: Baseline, 8 weeks
Population: A subset of randomized participants, who were >= 65 years of age and had ABPM measurements at both baseline and week 8, were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | VAL + AHU 400 mg | VAL + AHU 200 mg | VAL + AHU 100 mg | VAL + AHU 50 mg | VAL 320 mg | LCZ 400 mg | Placebo
Number analyzed (Participants) | 50 | 48 | 46 | 48 | 49 | 42 | 20
mmHg
  maSBP | -12.10 (1.04) | -16.08 (1.03) | -14.20 (1.08) | -12.25 (1.04) | -9.73 (1.02) | -11.88 (1.10) | -1.95 (1.59)
  maDBP | -4.94 (0.58) | -6.00 (0.57) | -4.86 (0.60) | -4.93 (0.58) | -4.58 (0.56) | -5.04 (0.61) | -0.01 (0.88)

14. Secondary Outcome: Number of Participants Who Achieved Blood Pressure Control and Blood Pressure Response
Description: Sitting BP measurements were performed at trough (23-26 hours post-morning dose). Blood pressure control was defined as msSBP/MSDBP < 140/90 mmHg. Blood pressure response in msSBP was defined as <140 mmHg or a reduction >= 20mmHg from baseline. Blood pressure response in msDBP was defined as < 90 mmHg or a reduction >= 10 mmHg from baseline.
Time Frame: 8 weeks
Population: Only participants of the full analysuis set (FAS), who had week 8 measurements, were included in the analysis. The FAS included all randomized participants who received at least one dose of double-blind study medication.
Measure: Number; unit: Number of participants
Arm/Group | VAL + AHU 400 mg | VAL + AHU 200 mg | VAL + AHU 100 mg | VAL + AHU 50 mg | VAL 320 mg | LCZ 400 mg | Placebo
Number analyzed (Participants) | 143 | 144 | 141 | 132 | 143 | 142 | 57
Number of participants
  Blood pressure control | 72 | 86 | 71 | 58 | 57 | 76 | 8
  msSBP response | 88 | 101 | 93 | 81 | 72 | 94 | 11
  msDBP response | 112 | 126 | 114 | 101 | 111 | 118 | 39

15. Secondary Outcome: Number of Participants With Adverse Events, Serious Adverse Events and Death
Description: Adverse event monitoring was conducted throughout the study.
Time Frame: 8 weeks
Population: Safety Analysis Set: The safety analysis set included all randomized participants who received at least one dose of study medication.
Measure: Number; unit: Number of participants
Arm/Group | VAL + AHU 400 mg | VAL + AHU 200 mg | VAL + AHU 100 mg | VAL + AHU 50 mg | VAL 320 mg | LCZ 400 mg | Placebo
Number analyzed (Participants) | 143 | 145 | 141 | 133 | 143 | 142 | 58
Number of participants
  Adverse events (non-serious and serious) | 40 | 31 | 29 | 25 | 38 | 42 | 20
  Serious adverse events | 3 | 1 | 1 | 0 | 1 | 1 | 1
  Deaths | 1 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | VAL + AHU 400 mg | VAL + AHU 200 mg | VAL + AHU 100 mg | VAL + AHU 50 mg | VAL 320 mg | LCZ 400 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 3/143 | 1/145 | 1/141 | 0/133 | 1/143 | 1/142 | 1/58
Other Adverse Events (participants affected / at risk) | 1/143 | 2/145 | 1/141 | 2/133 | 4/143 | 1/142 | 3/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VAL + AHU 400 mg (N=143) | VAL + AHU 200 mg (N=145) | VAL + AHU 100 mg (N=141) | VAL + AHU 50 mg (N=133) | VAL 320 mg (N=143) | LCZ 400 mg (N=142) | Placebo (N=58)
Sudden death (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Schizophrenia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VAL + AHU 400 mg (N=143) | VAL + AHU 200 mg (N=145) | VAL + AHU 100 mg (N=141) | VAL + AHU 50 mg (N=133) | VAL 320 mg (N=143) | LCZ 400 mg (N=142) | Placebo (N=58)
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 1 | 2 | 4 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.